CLINICAL TRIAL: NCT01633216
Title: Assessment of the Immunogenicity of Three Doses of Bivalent, Trivalent or Type One Monovalent Oral Poliovirus Vaccines Provided at 2 or 4 Week Intervals
Brief Title: Poliovirus Vaccine Trial in Bangladesh
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PR-11064
Record Dates: First submitted 2012-06-30; First posted 2012-07-04 (Estimated); Last update posted 2013-01-08 (Estimated); Status verified 2012-06

CONDITIONS: Healthy Infants
Keywords: poliovirus,; trivalent oral polio vaccine,; bivalent oral polio vaccine,; monovalent oral polio vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Bivalent OPV 2 week interval (Active Comparator): Group A will receive 3 doses of bOPV at 6, 8 and 10 weeks of age (2-week interval between doses).
  Interventions: Biological: Bivalent OPV 2 week interval
- Bivalent OPV 4 week interval (Active Comparator): Group B will receive 3 doses of bOPV at 6, 10 and 14 weeks of age (4-week interval between doses).
  Interventions: Biological: Bivalent OPV 4 week interval
- Monovalent OPV 2week interval (Active Comparator): Group C will receive 3 doses of mOPV1 at 6, 8 and 10 weeks of age (2-week interval between doses).
  Interventions: Biological: Monovalent OPV 2 week interval
- Monovalent OPV 4 week interval (Active Comparator): Group D will receive 3 doses of mOPV1 at 6, 10 and 14 weeks of age (4-week interval between doses).
  Interventions: Biological: Monovalent OPV 4 week interval
- Trivalent OPV 4 week interval (Active Comparator): Group E will receive 3 doses of tOPV at 6, 10 and 14 weeks of age (4-week interval between doses and similar to the current routine immunization schedule).
  Interventions: Biological: Trivalent OPV 4 week interval

INTERVENTIONS:
Biological: Bivalent OPV 2 week interval — Group A will receive 3 doses of bOPV at 6, 8 and 10 weeks of age (2-week interval between doses).
  Arms: Bivalent OPV 2 week interval
Biological: Bivalent OPV 4 week interval — Group B will receive 3 doses of bOPV at 6, 10 and 14 weeks of age (4-week interval between doses).
  Arms: Bivalent OPV 4 week interval
Biological: Monovalent OPV 2 week interval — Group C will receive 3 doses of mOPV1 at 6, 8 and 10 weeks of age (2-week interval between doses).
  Arms: Monovalent OPV 2week interval
Biological: Monovalent OPV 4 week interval — Group D will receive 3 doses of mOPV1 at 6, 10 and 14 weeks of age (4-week interval between doses).
  Arms: Monovalent OPV 4 week interval
Biological: Trivalent OPV 4 week interval — Group E will receive 3 doses of tOPV at 6, 10 and 14 weeks of age (4-week interval between doses and similar to the current routine immunization schedule).
  Arms: Trivalent OPV 4 week interval

SUMMARY:
This randomized clinical trial will assess the immune response in infants following administration of three types of oral poliovirus vaccine trivalent OPV (tOPV), monovalent OPV type 1 (mOPV1), bivalent OPV types 1 and 3 (bOPV) using two different schedules: a short schedule with administration at two week intervals and the usual schedule at four week intervals. The results of this study will guide the Global Polio Eradication Program in the implementation of new strategies that may: 1) improve the quality of the response to outbreaks following importation of wild poliovirus type 1 by shortening the interval at which several OPV doses are provided; 2) prevent alternate outbreaks of type 1 and type 3 poliovirus by using bOPV in outbreak responses in countries with weak routine immunization systems; and 3) prevent the emergence of type 2 vaccine-derived poliovirus through the replacement of tOPV with bOPV in immunization campaigns and routine immunization programs.

DETAILED DESCRIPTION:
This is a phase IV, randomized controlled clinical trial of three types of oral poliovirus vaccines provided at 2-week or 4-week intervals.

The study will enroll 1,000 participants from rural Matlab and urban Dhaka.

In this study infants will be given two different types of oral poliovirus vaccine, monovalent OPV type 1 (mOPV1) and bivalent OPV types 1 and 3 (bOPV) using two different schedules: a short schedule with administration at two week intervals and the usual schedule at four week intervals. The immune responses to these vaccines and schedules will be compared with the response to the routine oral polio vaccine schedule in Bangladesh of trivalent oral polio vaccine (tOPV) given at 4 week intervals.

The study will use a randomized controlled trial design. Eligible infants will be randomized at 6 weeks of age to one of five study arms: A) 3 doses of bOPV at 6, 8 and 10 weeks of age (2-week interval between doses); B) 3 doses of bOPV at 6, 10 and 14 weeks of age (4-week interval between doses); C) 3 doses of mOPV1 at 6, 8 and 10 weeks of age (2-week interval between doses); D) 3 doses of mOPV1 at 6, 10 and 14 weeks of age (4-week interval between doses); and E) 3 doses of tOPV at 6, 10 and 14 weeks of age (4-week interval between doses). Currently, tOPV is provided in routine immunization in Bangladesh at the same age as proposed in this study. bOPV, mOPV1 and mOPV3 are licensed in several countries and the World Health Organization (WHO) has recommended its use in immunization campaigns among children 0 to 5 years in response to circulation of type 1 and type 3 wild poliovirus, and to prevent outbreaks in countries at risk.

To assess the immunogenicity of each study vaccine and vaccination schedule, antibody titers against poliovirus types 1, 2 and 3 will be determined in sera extracted from blood collected before (at 6 weeks of age) and after receiving 3 doses of study vaccine. Seroconversion will be defined as a titer 4-fold higher than the expected fall in maternally derived antibodies, assuming a half life of 28 days. The initial antibody titer at 6 weeks of age will be used as the starting point for the expected decline in maternal antibody. We will calculate a one-sided 95% confidence interval for the difference between the proportion of seroconversions achieved in the short interval study arms and the longer interval study arms. If the confidence interval does not include 10%, we will conclude that the short interval is not inferior to the longer interval. This same analysis will be applied to the difference between bOPV and mOPV1.

This study will answer the following questions:

1. Is the immunogenicity of 3 doses of bOPV non inferior to that of 3 doses of mOPV1 against type 1 poliovirus?
2. Is an interval of 2 weeks between bOPV or mOPV1 doses non inferior to an interval of 4 weeks?
3. Will replacement of tOPV with bOPV in the routine immunization schedule achieve similar or higher proportions of children immune to type 1 and 3 polioviruses? The answers to these questions will guide the Global Polio Eradication Program in implementing new strategies that may: 1) improve the quality of the response to outbreaks following importation of wild poliovirus type 1 by shortening the interval at which several OPV doses are provided; and 2) prevent alternate outbreaks of type 1 and type 3 poliovirus by using bOPV instead of monovalent OPVs; and 3) prevent the emergence of type 2 vaccine-derived poliovirus through the replacement of tOPV with bOPVin immunization campaigns and in routine immunization programs.

ELIGIBILITY:
Inclusion Criteria:

* Healthy infants of 6 weeks of age (±2 days).
* Study families reside within the Health and Demographic Surveillance System (HDSS) area, service area of the ICDDR,B.
* Family able to understand and comply with planned study procedures

Exclusion Criteria:

* Family residence outside the ICDDR,B HDSS service area, or families expecting to move away during the study period, will be excluded.
* A diagnosis or suspicion of immunodeficiency disorder (either in the infant or in a member of the immediate family).
* A diagnosis or suspicion of bleeding disorder that would contraindicate venipuncture.
* Acute diarrhea, infection or illness at the time of the first visit (6 weeks of age) that would require infant's admission to a hospital or would contraindicate provision of OPV per country guidelines.
* Acute vomiting and intolerance to liquids within 24 hours before the first visit (6 weeks of age).
* Receipt of OPV or IPV at any time before enrollment based upon mother's recall or immunization card if available.
* Because of contact transmission of vaccine poliovirus strains, newborns from multiple births will be excluded from the study to prevent transmission of vaccine strains received during routine immunization from the twin to the study participant.

Ages: 6 Weeks to 6 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1000 (Actual)
Dates: Start 2012-05; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Immunogenicity | 7 months
  To assess the immunogenicity of each study vaccine and vaccination schedule, antibody titers against poliovirus types 1, 2 and 3 will be determined in sera extracted from blood collected before (at 6 weeks of age) and after receiving 3 doses of study vaccine.

CONTACTS AND LOCATIONS:
Locations (2):
- Bangladesh (2):
  - Matlab, Matlab, Chandpur
  - Mirpur, Dhaka, Dhaka Division

REFERENCES:
- [Derived] Emperador DM, Velasquez DE, Estivariz CF, Lopman B, Jiang B, Parashar U, Anand A, Zaman K. Interference of Monovalent, Bivalent, and Trivalent Oral Poliovirus Vaccines on Monovalent Rotavirus Vaccine Immunogenicity in Rural Bangladesh. Clin Infect Dis. 2016 Jan 15;62(2):150-6. doi: 10.1093/cid/civ807. Epub 2015 Sep 8. PMID 26349548
- [Derived] Estivariz CF, Anand A, Gary HE Jr, Rahman M, Islam J, Bari TI, Wassilak SG, Chu SY, Weldon WC, Pallansch MA, Heffelfinger JD, Luby SP, Zaman K. Immunogenicity of three doses of bivalent, trivalent, or type 1 monovalent oral poliovirus vaccines with a 2 week interval between doses in Bangladesh: an open-label, non-inferiority, randomised, controlled trial. Lancet Infect Dis. 2015 Aug;15(8):898-904. doi: 10.1016/S1473-3099(15)00094-8. Epub 2015 Jun 17. PMID 26093980